CLINICAL TRIAL: NCT02347709
Title: Differential Clinical, Molecular, and Pathological Characteristics of Neuropathy in Type 2 Diabetics With and Without Lower Extremity Wounds-a Pilot Study
Brief Title: Differential Characteristics of Neuropathy in Type 2 Diabetics With and Without Lower Extremity Wounds
Status: Withdrawn | Type: Observational
Why Stopped: PI departure
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 14024
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2015-12

CONDITIONS: Diabetic Foot Ulcer; Diabetic Neuropathy; Type 2 Diabetes
Keywords: Diabetic Foot Ulcer; DFU; Type 2 Diabetes; Neuropathy
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies; Diabetes Mellitus, Type 2 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue samples will be obtained via 3mm punch biopsy during standard of care wound debridement.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1/Diabetic Foot Ulcer: Group 1 will be recruited from the Wound Center, and will include patients with a diagnosis of Type 2 Diabetes (defined as HgA1c ≥5.9%), and a diabetic foot ulcer (defined as a break in the skin on the foot). Subjects in this group will complete a survey, undergo a Comprehensive Neuropathy Evaluation, and have a photograph and biopsy of their Diabetic Foot Ulcer in addition to the standard of care.
  Interventions: Procedure: Diabetic Foot Ulcer Biopsy; Other: Survey; Other: Comprehensive Neuropathy Assessment; Other: Wound Photography
- Group 2/Diabetic Neuropathy: Group 2 will be recruited from the Neurology clinic and will include patients with a diagnosis of Type 2 Diabetes (defined as HgA1c ≥ 5.9%) and neuropathy. Subjects in this group will complete a survey and undergo a Comprehensive Neuropathy Evaluation in addition to the standard of care.
  Interventions: Other: Survey; Other: Comprehensive Neuropathy Assessment
- Group 3/Type 2 Diabetes: Group 3 will be recruited from the Endocrinology clinic and will include patients with a diagnosis of Type 2 Diabetes (defined as HgA1c ≥ 5.9%) who currently do not have a diagnosis of neuropathy or a diabetic foot ulcer. Subjects in this group will complete a survey and undergo a Comprehensive Neuropathy Evaluation in addition to the standard of care.
  Interventions: Other: Survey; Other: Comprehensive Neuropathy Assessment

INTERVENTIONS:
Procedure: Diabetic Foot Ulcer Biopsy — Specimens from both the wound edge and a distal area of skin of patients will be obtained via 3 mm punch biopsy in the Winthrop University Hospital Wound Care Center. Biopsies will be collected from the wound edge prior to routine debridement using the following standard procedures, including the use of anesthetic if needed.
  Groups: Group 1/Diabetic Foot Ulcer
Other: Survey — Study subjects from all three groups will be asked to complete a one-page Focused Neuropathy Evaluation. Providers will complete a one-page Focused Neuropathy Evaluation and a complete neurological examination and sensation assessment.
Other: Comprehensive Neuropathy Assessment — Standard Monofilament Exam, Vibration Assessment, and Temperature Assessment will be performed on all patients in all study groups.
Other: Wound Photography — Digital photographs and wound measurements for patients in Study Group 1 will be obtained per standard protocol at baseline and all subsequent visits.
  Groups: Group 1/Diabetic Foot Ulcer

SUMMARY:
The primary purpose of this study is to determine the degree of loss of epidermal nerve fibers near a foot wound in patients with diabetic foot ulcers. The secondary purpose will be to determine whether the degree of epidermal nerve fiber loss, the clinical examination, nerve conduction studies or the molecular profile correlates with appearance of lower extremity ulcers in patients with diabetes.

DETAILED DESCRIPTION:
Neuropathy is a common complication of diabetes seen in up to 43% of patients with diabetes. The relationship between neuropathy and diabetic lower extremity wounds is strong and in fact, 80% of patients with an existing diabetic foot ulcer (DFU) have neuropathy. Understanding the factors that contribute to the increased risk of wounds in patients with neuropathy is important in creating optimal strategies to reduce this risk.

Traditionally, the severity of diabetic neuropathy has been evaluated using the clinical exam and nerve conduction studies. More recently, new techniques such as intra-epidermal nerve fiber density have shown promise in evaluating neuropathy especially the small nerve fiber neuropathies that might affect pain sensation and autonomic function. There are also new molecular markers that may correlate with the risk of neuropathy that may also be useful in clinically evaluating the diabetic patient with neuropathy.

The primary purpose of this study is to determine the degree of loss of epidermal nerve fibers near a foot wound in patients with diabetic foot ulcers. The secondary purpose will be to determine whether the degree of epidermal nerve fiber loss, the clinical examination, nerve conduction studies or the molecular profile correlates with appearance of lower extremity ulcers in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Type 2 Diabetes defined as HgA1c ≥ 5.9%
* Must be willing and able to provide written Informed Consent

Exclusion Criteria:

* Active osteomyelitis
* Gangrene
* Purulent drainage
* Any experimental drugs applied topically or taken by mouth within 4 weeks of study entry
* INR > 2.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include eligible patients from three Winthrop outpatient services, separated into three study groups. Based on demographic data from this institution, we expect our population sample to be representative of all major races and ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Measure the degree of loss of epidermal nerve fibers near a lower extremity diabetic wound using Intra-epidermal Nerve Fiber Density analysis. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stecker, MD, PhD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States